CLINICAL TRIAL: NCT07314515
Title: The ECHO Study: Compassion-focused Therapy for Young Voice Hearers and Their Caregivers
Acronym: ECHO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Region Syddanmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1852876
Record Dates: First submitted 2025-12-03; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Hallucinations, Auditory
Keywords: voice hearing
MeSH Terms: conditions — Hallucinations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 10 sessions manualized CFT treatment for young voice heares (Experimental): 60 voice hearing patients age 13-18 years old 20 patients with first-episode schizophrenia age 18-21
  Interventions: Behavioral: ECHO Manualized CFT treatment for young voice heares

INTERVENTIONS:
Behavioral: ECHO Manualized CFT treatment for young voice heares — A manualized 10 session, intervention inspired by compassion focused therapy. A primary caretaker paticipates in 5 sessions.
  Other Names: Data is collected 3 months prior to CFT treatment, immediately before the start of treatment, immediately after treatment is completed, and at 1 month follow-up

SUMMARY:
In this project, a 10-session treatment program was developed aimed at young people who experience voice hearing. The treatment has potential to easily be implemented in everyday clinical practice in Child and Adolescent Psychiatry, and eventually in Educational Psychological Counselling (PPR) and the newly established STIME services (low-threshold municipal treatment offers for children and young people).

As part of the treatment, the young person's caregivers are involved. This means a high degree of involvement from adults who know the young person well and are part of their daily life.

In addition to traditional Compassion-focuced therapy (CFT), the treatment is expanded with an intervention where an audio file is recorded with content corresponding to the adolescent's voice hearing. The parents are invited to listen to the audio file while participating in a therapy session. This will help improve the caregivers understanding of the young person's experiences and challenges.

ELIGIBILITY:
Inclusion Criteria:

* The participants should have been referred to a child and adolescent psychiatric hospital in Denmark .
* The participants have heard voices within the last 2 weeks.
* The participant can hear the content of the voices. The content takes the form of spoken works.
* A caregiver who can participate in 5 sessions

Exclusion Criteria:

* Participants has an estimated IQ under 70
* Participants who don't speak and understand Danish,
* Current drug misuse / abuse (during sessions)
* Brain injury or neurological disorder e.g. severe epilepsy
* Impaired vision or hearing to a degree that makes participation in therapy under normal conditions impossible.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Interpretation and relationship with the voices | Data is collected 3 months prior to CFT treatment, immediately before the start of treatment, immediately after treatment is completed, and at 1 month follow-up.
  Psychotic symptoms are measured with: BAVQ-R (Beliefs about Voices Questionnaire - Revised) (Chadwick et al., 2000).( 35 items are rated (0-3) total minimum score 0, maximum score 105. Some scores indicate higher distress, while other indicate lower distress).
Severity and phenomenological characteristics of voice hearing | Data is collected 3 months prior to CFT treatment, immediately before the start of treatment, immediately after treatment is completed, and at 1 month follow-up.
  PSYRATS AH (Psychotic Symptoms Rating Scale Auditory Hallucinations) (Haddock et al., 1999). (11 items are rated (0-4) total minimum score 0, maximum score 44. Higher score being more severe)
Perceived ability to control or influence the voices | Data is collected 3 months prior to CFT treatment, immediately before the start of treatment, immediately after treatment is completed, and at 1 month follow-up.
  The Yale Control Over Perceptual Experiences (COPE) Scales measures voluntary control over voices such as being able to intentionally influence the timing, frequency, or intensity of voice hearing experiences (Mourgues et al., 2022). (36 items are rated (1-7) total minimum score 36, maximum score 252. Higher scores indicate stronger perceived control over voices)

SECONDARY OUTCOMES:
Social Cognition | Social cognition is tested 3 months before treatment and right after
  Social cognition is tested with TASIT 2A DK (The Awareness of Social Inference Test) (McDonald et al., 2003). (60 items are rated, minimum total score 0, maximum score is 60. Lower score being more severe)
Subjective experience of feeling safe, accepted, and soothed in social relationships. | Data is collected 3 months prior to CFT treatment, immediately before the start of treatment, immediately after treatment is completed, and at 1 month follow-up
  SSPS (Social safeness and pleasure scale) (Gilbert et al., 2009). (11 items are rated (1-5). Total minimum 11, total maximum 55. Lower score being more severe).
Compassion towards self. | Data is collected 3 months prior to CFT treatment, immediately before the start of treatment, immediately after treatment is completed, and at 1 month follow-up
  SCS-SF (Self-Compassion Scale Short Form) (Raes et al., 2011; Neff et al., 2019) (12 items are rated (1-5) total minimum 12, total maximum 60. Lower score being more severe).
Subjective sense of interpersonal closeness and belonging | Data is collected 3 months prior to CFT treatment, immediately before the start of treatment, immediately after treatment is completed, and at 1 month follow-up
  The Social Connectedness Scale Revised (Lee et al., 1995; Sabitelli et al., 2005). (8 items are rated (1-6). Total minimum score 8, total maximum score 48. Lower score being more severe).
Perceived availability and adequacy of social support | Data is collected 3 months prior to CFT treatment, immediately before the start of treatment, immediately after treatment is completed, and at 1 month follow-up
  MSPSS (The Multidimensional Scale of Perceived Social Support) (Zimet et al. 1988).(12 items are rated (1-7) total minimum 12, total maximum 84. Lower score being more severe).

OTHER OUTCOMES:
Primary caregivers | Before treatment
  Factual information about the young person: Education, cohabiting or divorced parents, the young person's residence, family history of mental illness, diagnosis and medication of the young person
Additional questions | Data is collected 3 months prior to CFT treatment, immediately before the start of treatment, immediately after treatment is completed, and at 1 month follow-up
  Additionally, questions are asked about how well you feel your parents understand you (e.g., do they know what motivates you and what scares you?) (Likert scale 1-10). Questions about daily stress, sleep, violence and abuse, well-being and quality of life, interaction with family and friends (from the "How are you?" survey among youth in the Central Denmark Region). Quality of life is measured with WHO-5.

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Heriot-Maitland, Dr., Study Chair — Balanced Minds
Locations (1):
- Psychiatriatric Children and Youth Hospital, Esbjerg, Denmark

REFERENCES:
- [Background] Heriot-Maitland C. Position paper - CFT for psychosis. Psychol Psychother. 2024 Mar;97(1):59-73. doi: 10.1111/papt.12490. Epub 2023 Aug 14. PMID 37578215
- [Result] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Result] Neff KD, Toth-Kiraly I, Yarnell LM, Arimitsu K, Castilho P, Ghorbani N, Guo HX, Hirsch JK, Hupfeld J, Hutz CS, Kotsou I, Lee WK, Montero-Marin J, Sirois FM, de Souza LK, Svendsen JL, Wilkinson RB, Mantzios M. Examining the factor structure of the Self-Compassion Scale in 20 diverse samples: Support for use of a total score and six subscale scores. Psychol Assess. 2019 Jan;31(1):27-45. doi: 10.1037/pas0000629. Epub 2018 Aug 20. PMID 30124303
- [Result] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Result] Gilbert, P., Introducing compassion-focused therapy. Advances in psychiatric treatment, 2009. 15(3): p. 199-208.
- [Result] Mourgues C, Hammer A, Fisher V, Kafadar E, Quagan B, Bien C, Jaeger H, Thomas R, Sibarium E, Negreira AM, Sarisik E, Polisetty V, Nur Eken H, Imtiaz A, Niles H, Sheldon AD, Powers AR. Measuring Voluntary Control Over Hallucinations: The Yale Control Over Perceptual Experiences (COPE) Scales. Schizophr Bull. 2022 May 7;48(3):673-683. doi: 10.1093/schbul/sbab144. PMID 35089361
- [Result] Woods, S. W., Parker, S., Kerr, M. J., Walsh, B. C., Wijtenburg, S. A., Prunier, N., Nunez, A. R., Buccilli, K., Mourgues-Codern, C., Brummitt, K., Kinney, K. S., Trankler, C., Szacilo, J., Colton, B.-L., Ali, M., Haidar, A., Billah, T., Huynh, K., Ahmed, U., Adery, L. L., Marcy, P. J., Allott, K., Amminger, P., Arango, C., Broome, M. R., Cadenhead, K. S., Chen, E. Y. H., Choi, J., Conus, P., Cornblatt, B. A., Glenthøj, L. B., Horton, L. E., Kambeitz, J., Kapur, T., Keshavan, M. S., Koutsouleris, N., Langbein, K., Lavoie, S., Diaz-Caneja, C. M., Mathalon, D. H., Mittal, V. A., Nordentoft, M., Pasternak, O., Pearlson, G. D., Gaspar, P. A., Shah, J. L., Smesny, S., Stone, W. S., Strauss, G. P., Wang, J., Corcoran, C. M., Perkins, D. O., Schiffman, J., Perez, J., Mamah, D., Ellman, L. M., Powers, A. R. III, Coleman, M. J., Anticevic, A., Fusar-Poli, P., Kane, J. M., Kahn, R. S., McGorry, P. D., Bearden, C . E., Shenton, M. E., Nelson, B., Calkins, M. E., Hendricks, L., Bouix, S., Addington, J., McGlashan, T. H., Yung, A. R., & The Accelerating Medicines Partnership Schizophrenia (2024). Development of the PSYCHS: Positive SYmptoms and Diagnostic Criteria for the CAARMS Harmonized with the SIPS. Early Intervention in Psychiatry, 18(4), 255-272. https://doi.org/10.1111/eip.13457
- [Result] Chandwick P, Lees S, Birchwood M. The revised Beliefs About Voices Questionnaire (BAVQ-R). Br J Psychiatry. 2000 Sep;177:229-32. doi: 10.1192/bjp.177.3.229. PMID 11040883
- [Result] McDonald S, Flanagan S, Rollins J, Kinch J. TASIT: A new clinical tool for assessing social perception after traumatic brain injury. J Head Trauma Rehabil. 2003 May-Jun;18(3):219-38. doi: 10.1097/00001199-200305000-00001. PMID 12802165